CLINICAL TRIAL: NCT04126031
Title: A PHASE 2A, 2-PART, OPEN-LABEL, NON-RANDOMIZED, MULTICENTER, SINGLE AND MULTIPLE DOSE TRIAL TO EVALUATE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF CEFTAZIDIME AND AVIBACTAM IN NEONATES AND INFANTS FROM BIRTH TO LESS THAN 3 MONTHS OF AGE WITH SUSPECTED OR CONFIRMED INFECTIONS DUE TO GRAM-NEGATIVE PATHOGENS REQUIRING INTRAVENOUS ANTIBIOTIC TREATMENT
Brief Title: Evaluation of Pharmacokinetics, Safety, and Tolerability of Ceftazidime-avibactam in Neonates and Infants.
Acronym: NOOR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following regulatory consultation, the Sponsor has decided to terminate the study and analyze the current dataset. The decision to terminate was solely based on a business decision, not due to safety concerns.
Sponsor: Pfizer (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C3591024; 2018-002800-16 (EudraCT Number); NOOR (Other: Alias Study Number)
Record Dates: First submitted 2019-09-27; First posted 2019-10-14 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Gram-negative Bacterial Infection
Keywords: Gram-negative, ceftazidime-avibactam, neonate, infant
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Intervention Model Description: Non-randomized, 2-part with three age cohorts in each part
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A, Cohorts 1-3 (Experimental): Single dose pharmacokinetics. This arm will include three age cohorts.
  Interventions: Drug: Part A: Single Dose Ceftazidime-Avibactam, Cohorts 1-3
- Part B, Cohorts 1-3 (Experimental): Multi-dose pharmacokinetics. This arm will include three age cohorts.
  Interventions: Drug: Part B: Multiple-dose Ceftazidime-Avibactam, Cohorts 1-3

INTERVENTIONS:
Drug: Part A: Single Dose Ceftazidime-Avibactam, Cohorts 1-3 — Single intravenous infusion of ceftazidime-avibactam over 2 hours
  Arms: Part A, Cohorts 1-3
Drug: Part B: Multiple-dose Ceftazidime-Avibactam, Cohorts 1-3 — Multiple intravenous infusions of ceftazidime-avibactam over 2 hours, repeated every 8 hours up to 14 days
  Arms: Part B, Cohorts 1-3

SUMMARY:
This study will assess the pharmacokinetics, safety, and tolerability of single and multiple doses of intravenous ceftazidime-avibactam in hospitalized infants and neonates from 26 weeks gestation to 3 months of age. In Part A of the study all patients will receive a single dose of ceftazidime-avibactam. In Part B all patients will received multiple doses of ceftazidime-avibactam. Efficacy will be assessed in the infants and neonates receiving multiple doses of ceftazidime-avibactam.

DETAILED DESCRIPTION:
This is a 2-part, Phase 2a, non-randomized, open-label multicenter, multinational study of intravenous ceftazidime-avibactam in hospitalized neonates and infants with suspected or confirmed bacterial infection. In Part A of the study, patients already receiving intravenous antibacterial therapy with another antibiotic will receive a single intravenous dose of ceftazidime-avibactam followed by observation for 48 hours and a Late Follow-Up assessment 4-5 weeks later. In Part B of the study, patients with suspected or confirmed Gram-negative bacterial infections requiring intravenous antibacterial therapy will receive multiple doses of intravenous ceftazidime-avibactam for up to 14 days. At the discretion of the investigator, patients may also receive other antibiotics if the infection is suspected to include Gram-positive bacteria, multi-drug resistant Gram-negative bacteria, or anaerobic bacteria. At the discretion of the investigator, patients may be switched to oral therapy or outpatient parenteral antimicrobial therapy with an alternative antibiotic after receiving intravenous ceftazidime-avibactam for at least 48 yhours. Clinical outcomes will be assessed at the End of Intravenous (EOIV) treatment with ceftazidime-avibactam, the End-of-Therapy (EOT), the Test-of-Cure (TOC) at 7-14 days after the last study therapy and at a Late Follow-Up (LFU) visit, 28-55 days after the last dose of ceftazidime-avibactam. Safety assessments will occur throughout the study. Ceftazidime-avibactam blood levels will be assessed during the first 12 hours after the single dose of ceftazidime-avibactam in Part A and during 12 hours after at least 3 consecutive doses of ceftazidime-avibactam in Part B.

ELIGIBILITY:
Inclusion Criteria (All Subjects):

1. Evidence of a personally signed and dated informed consent document indicating that the subject's parent(s), legal guardian, or legally acceptable representative has been informed of all pertinent aspects of the study.
2. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Male or female neonates and infants with age at Screening:

Cohort 1: Full term infants (gestational age ≥ 37 weeks) with chronological age >28 days to <3 months (<89 days) or pre-term infants with corrected age >28 days to <3 months (<89 days). A maximum of 3 pre-term corrected age infants may be enrolled in each part (A and B) of Cohort 1. Sites will be notified in writing if this limit is reached.

Cohort 2: Full term neonates (gestational age ≥ 37 weeks) from birth to ≤ 28 days.

Cohort 3: Pre-term neonates (gestational age ≥ 26 to <37 weeks) from birth to ≤ 28 days.

Corrected age = Subtract the number of weeks born before 40 weeks of gestation from the chronological age.

Inclusion Criteria for Part A Subjects Only:

1. Hospitalized and receiving intravenous antibacterial therapy for the treatment of a suspected or confirmed bacterial infection.

Inclusion Criteria for Part B Subjects Only:

1. Hospitalized with suspected or confirmed aerobic Gram-negative bacterial infection requiring intravenous antibacterial therapy.
2. Subjects must meet at least 1 clinical and 1 laboratory criterion or meet at least 2 of the clinical criteria:

Clinical Criteria:

1. Hypothermia (<36ºC) OR fever (>38.5ºC);
2. Bradycardia OR tachycardia OR rhythm instability;
3. Urine output 0.5 to 1 mL/kg/h OR hypotension OR mottled skin OR impaired peripheral perfusion;
4. Petechial rash OR sclerema neonatorum;
5. New onset or worsening of apnea episodes OR tachypnea episodes OR increased oxygen requirements OR requirement for ventilation support;
6. Feeding intolerance OR poor suckling OR abdominal distension;
7. Irritability;
8. Lethargy;
9. Hypotonia.

Laboratory Criteria:

1. White blood cell count ≤ 4.0 × 10^9/L OR ≥ 20.0 × 10^9/L;
2. Immature to total neutrophil ratio >0.2;
3. Platelet count ≤ 100 × 10^9/L;
4. C reactive protein (CRP) >15 mg/L OR procalcitonin ≥ 2 ng/mL;
5. Hyperglycemia OR Hypoglycemia;
6. Metabolic acidosis.

Exclusion Criteria (All Subjects):

1. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
2. Participation in another clinical study involving investigational drug(s) within 30 days prior to study entry and/or during this study participation or have previously participated in the current study or in another study of CAZ-AVI (in which an active agent was received).
3. Use of potent inhibitors of organic anion transporters OAT1 and/or OAT3 (eg, probenecid, p-aminohippuric acid (PAH), or teriflunomide) are prohibited. This prohibition of OAT1 and/or OAT3 inhibitors also applies to the mothers of any neonates or infants who are breast feeding during the trial.
4. Other acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
5. Documented history of any hypersensitivity or allergic reaction to any beta-lactam antibiotic.
6. Refractory septic shock within 24 hours before screening that does not resolve after 60 minutes of vasopressor therapy.
7. Moderate or severe renal impairment defined as serum creatinine ≥ 2 times the upper limit of normal (ULN) for age OR urine output <0.5 mL/kg/h (measured over at least 8 hours) OR requirement for dialysis. Deterioration of renal function after enrollment during Part B of the study will be handled on a case-by-case basis in discussion with the Medical Monitor.
8. Evidence of progressively fatal underlying disease, or life expectancy of ≤ 60 days.
9. Documented history of seizure.
10. Active acute viral hepatitis or acute hepatic failure.
11. Known Clostridium difficile associated diarrhea.
12. Requiring or currently taking antiretroviral therapy for human immunodeficiency virus (HIV) or known HIV positive mother.
13. Any condition (eg, cystic fibrosis, urea cycle disorders), antepartum/peripartum factors, or procedures that would, in the opinion of the Investigator, make the subject unsuitable for the study, place a subject at risk, or compromise the quality of data.
14. Treatment with ceftazidime within 12 hours of CAZ-AVI administration.

Exclusion Criteria for Part A Subjects Only:

1. Subject received a blood or a blood component transfusion within 24 hours of the start of CAZ AVI infusion.
2. Subject is expected to be discharged less than 24 hours after the start of CAZ AVI infusion.

Exclusion Criteria for Part B Subjects Only:

1. At study entry, subject has confirmed or strongly suspected infection with a pathogen known to be resistant to CAZ-AVI or only a Gram-positive pathogen or viral, fungal, or parasitic pathogens as the sole cause of infection.
2. Confirmed or suspected central nervous system (CNS) infection (eg, meningitis, brain abscess, subdural abscess).
3. Anticipated need for antibacterial therapy longer than 14 days (eg, osteomyelitis, endocarditis). This applies to both study treatment with CAZ-AVI as well as adjunctive IV antibacterial treatment for suspected co infection with Gram-positive organisms or multi drug resistant Gram-negative organisms.
4. Receipt of more than 24 hours of nonstudy systemic antibacterial treatment for Gram-negative organisms after culture and before administration of study doses of CAZ-AVI. Empiric coverage with an aminoglycoside for suspected multidrug resistant organisms is permitted, provided CAZ-AVI is initiated within 24 hours after culture.
5. Intravenous treatment with chloramphenicol within 24 hours of administration of study doses of CAZ-AVI.
6. Subject is expected to be discharged less than 48 hours after the start of CAZ-AVI infusion.

Ages: 0 Days to 88 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (5):
  - Tufts Children's Hospital at Tufts Medical Center, Boston, Massachusetts
  - Duke University Investigational Drug Services, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Utah, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
- Tallinn Children's Hospital, Tallinn, Estonia
- Greece (3):
  - Athens General Children's Hospital "Panagioti and Aglaias Kyriakou", Athens, Ampelokipi
  - "ATTIKON" University General Hospital, Chaïdári, Athens
  - "Hippokration" General Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Kanizsai Dorottya Korhaz, Nagykanizsa
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Oktatókórház, Jósa András Oktatókórház, Nyíregyháza
- Kasturba Medical College and Hospital, Manipal, Karnataka, India
- Ospedale Pediatrico Bambino Gesu, Rome, RM, Italy
- Univerzitna nemocnica Martin, Martin, Slovakia
- Taiwan (3):
  - Hsinchu Mackay Memorial Hospital, Department of Pharmacy, Hsinchu, R.o.c
  - Hsinchu Mackay Memorial Hospital, Hsinchu
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Bradley J, Roilides E, Tawadrous M, Yan JL, Soto E, Stone GG, Kamat S, Irani P, England R. Pharmacokinetics and Safety of Ceftazidime-Avibactam in Neonates and Young Infants: A Phase 2a, Multicenter Prospective Trial. J Pediatric Infect Dis Soc. 2025 May 13;14(5):piaf028. doi: 10.1093/jpids/piaf028. PMID 40251980
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3591024

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 52 participants were screened, out of which 4 participants were screen failures and 48 were enrolled to the study. 27 participants in Part A and 21 participants in Part B.
Groups:
- Part A: Cohort 1: On Day 1 participants aged 28days to less than (<) 3 months old received a single intravenous (IV) infusion of ceftazidime-avibactam (CAZ-AVI) 30 milligrams per kilogram (mg/kg) CAZ and 7.5 mg/kg AVI over a 2-hour (+10 min) period.
- Part A: Cohort 2: On Day 1 participants aged greater than or equal to(>=) 37weeks and less than or equal to (<=) 28 days old received a single IV infusion of CAZ-AVI 20 mg/kg CAZ and 5.0 mg/kg AVI over a 2-hour (+10 min) period.
- Part A: Cohort 3: On Day 1 participants aged >=26 week to <37weeks and <=28days old received a single IV infusion of CAZ-AVI 20 mg/kg CAZ and 5.0 mg/kg AVI over a 2-hour (+10 min) period.
- Part B: Cohort 1: On Day 1 participants aged 28days to <3 months old received a single IV infusion of CAZ-AVI 30 milligrams per kilogram (mg/kg) CAZ and 7.5 mg/kg AVI over a 2-hour (+10 min) period every 8 hours (+1 hour).
- Part B: Cohort 2: On Day 1 participants aged >= 37weeks and <= 28days old received a single IV infusion of CAZ-AVI 20 mg/kg CAZ and 5.0 mg/kg AVI over 2-hour (+10 min) period every 8 hours (+1 hour).
- Part B: Cohort 3: On Day 1 participants aged >=26weeks to <37weeks and <=28days old received a single IV infusion of CAZ-AVI 20 mg/kg CAZ and 5.0 mg/kg AVI over a 2-hour (+10 min) period every 8 hours (+1 hour).
Period: Part A
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3 | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Started | 10 | 8 | 9 | 0 | 0 | 0
Treated | 9 | 8 | 8 | 0 | 0 | 0
Completed | 9 | 8 | 8 | 0 | 0 | 0
Not Completed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3 | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Started | 0 | 0 | 0 | 8 | 5 | 8
Completed | 0 | 0 | 0 | 8 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Pre-existing hypertransaminasemia | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis sets for Part A and Part B included participants who received any amount of the investigational drug (CAZ-AVI) in the respective part.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3 | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3 | Total
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 5 | 8 | 46
Age, Continuous [Mean (Standard Deviation); unit: Days] | 59.0 (15.73) | 19.3 (9.00) | 14.6 (7.46) | 51.1 (18.16) | 15.80 (7.63) | 17.8 (8.99) | 31.13 (22.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 3 | 1 | 6 | 25
  Male | 4 | 4 | 2 | 5 | 4 | 2 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 7 | 7 | 7 | 8 | 5 | 8 | 42
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 00 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 1 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2 | 0 | 0 | 4
  White | 6 | 5 | 7 | 5 | 5 | 8 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentrations of Ceftazidime and Avibactam 2 Hours Post-dose: Part A
Time Frame: 2 hours post dose on Day 1
Population: The Pharmacokinetic (PK) analysis set for Part A was defined as participants who received a single IV dose of CAZ-AVI in Part A.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3
Number analyzed (Participants) | 9 | 8 | 8
Nanogram per milliliter
  Ceftazidime | 104544.4 (113161.34) [lower limit 113161.34] | 35537.5 (13473.88) [lower limit 13473.88] | 53212.5 (25972.32) [lower limit 25972.32]
  Avibactam | 19210.0 (18747.86) [lower limit 18747.86] | 6910.0 (2553.50) [lower limit 2553.50] | 10570.0 (4342.69) [lower limit 4342.69]

2. Primary Outcome: Plasma Concentrations of Ceftazidime and Avibactam 2 Hours and 30 Minutes Post-dose: Part A
Time Frame: 2 hours and 30 minutes post dose on Day 1
Population: PK analysis set for Part A was defined as participants who received a single IV dose of CAZ-AVI in Part A. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3
Number analyzed (Participants) | 9 | 7 | 8
Nanogram per milliliter
  Ceftazidime | 76822.2 (106423.76) [lower limit 106423.76] | 32571.4 (10842.00) [lower limit 10842.00] | 49012.5 (18832.45) [lower limit 18832.45]
  Avibactam | 13250.0 (16906.67) [lower limit 16906.67] | 6251.4 (2363.99) [lower limit 2363.99] | 9788.8 (2956.39) [lower limit 2956.39]

3. Primary Outcome: Plasma Concentrations of Ceftazidime and Avibactam of 7 Hours Post-dose: Part A
Time Frame: 7 hours post dose on Day 1
Population: PK analysis set for Part A was defined as participants who received a single IV dose of CAZ-AVI in Part A.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3
Number analyzed (Participants) | 9 | 8 | 8
Nanogram per milliliter
  Ceftazidime | 15635.6 (15243.22) [lower limit 15243.22] | 8305.0 (6728.50) [lower limit 6728.50] | 17608.8 (8165.42) [lower limit 8165.42]
  Avibactam | 2058.2 (1670.32) [lower limit 1670.32] | 1190.4 (998.69) [lower limit 998.69] | 3475.6 (1931.10) [lower limit 1931.10]

4. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs): Part B
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in participant hospitalization; life-threatening experience (immediate risk of dying) ; persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Day 1 up to maximum of Day 49
Population: Safety analysis set for Part B included all participants who received any amount of the investigational drug (CAZ-AVI) in the Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 8 | 5 | 8
Participants
  AEs | 4 | 4 | 7
  SAEs | 1 | 2 | 2

5. Primary Outcome: Number of Participants Who Died: Part B
Time Frame: Day 1 up to maximum of Day 49
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 8 | 5 | 8
Participants | 0 | 0 | 1

6. Primary Outcome: Number of Participants Who Discontinued Treatment and Study Due to AEs: Part B
Time Frame: Day 1 up to maximum of Day 49
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 8 | 5 | 8
Participants
  Discontinued from study due to AEs | 0 | 0 | 2
  Discontinued study drug due to AE and continue study | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs): Part A
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Day 1 up to maximum of Day 35
Population: Safety analysis set for Part A included all participants who received any amount of the investigational drug (CAZ-AVI) in the Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3
Number analyzed (Participants) | 9 | 8 | 8
Participants
  AEs | 4 | 2 | 2
  SAEs | 2 | 0 | 1

8. Secondary Outcome: Number of Participants Who Died: Part A
Time Frame: Day 1 up to maximum of Day 35
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3
Number analyzed (Participants) | 9 | 8 | 8
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Discontinued Treatment and Study Due to AEs: Part A
Time Frame: Day 1 up to maximum of Day 35
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3
Number analyzed (Participants) | 9 | 8 | 8
Participants
  Discontinued from study due to AEs | 0 | 0 | 0
  Discontinued study drug due to AE and continue study | 0 | 0 | 0

10. Secondary Outcome: Plasma Concentrations of Ceftazidime and Avibactam 2 Hours, 2 Hours and 30 Minutes, 7 Hours Post Doses on Day 1: Part B
Time Frame: 2 hours, 2 hours 30 mins, and 7 hours post dose on Day 1
Population: PK analysis set for Part B was defined as participants who received at least 3 consecutive doses of CAZ-AVI in Part B. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 8 | 4 | 8
Nanograms per milliliter
  Ceftazidime: 2 hours | 52950.0 (17565.47) [lower limit 17565.47] | 48625.0 (17010.46) [lower limit 17010.46] | 43711.3 (22229.93) [lower limit 22229.93]
  Ceftazidime: 2 hours 30 mins | 43037.5 (17433.21) [lower limit 17433.21] | 39000.0 (4415.88) [lower limit 4415.88] | 42465.0 (26800.19) [lower limit 26800.19]
  Ceftazidime: 7 hours | 8323.8 (4805.65) [lower limit 4805.65] | 16735.0 (9070.87) [lower limit 9070.87] | 18658.4 (18268.92) [lower limit 18268.92]
  Avibactam: 2 hours | 10340.0 (3262.63) [lower limit 3262.63] | 11330.0 (2012.53) [lower limit 2012.53] | 9410.1 (5551.00) [lower limit 5551.00]
  Avibactam: 2 hours 30 mins | 6825.0 (2386.26) [lower limit 2386.26] | 9380.0 (2317.14) [lower limit 2317.14] | 9064.0 (5694.05) [lower limit 5694.05]
  Avibactam: 7 hours | 1025.3 (592.83) [lower limit 592.83] | 3787.5 (2533.46) [lower limit 2533.46] | 3890.5 (3867.47) [lower limit 3867.47]

11. Secondary Outcome: Number of Participants According to Clinical Outcome At End of IV Treatment(EOIV), End of Treatment(EOT), Test of Cure(TOC) and Late Follow-Up(LFU): Intent to Treat (ITT) Analysis Population: Part B
Description: Clinical outcome assessed based on clinical cure, improvement, failure, indeterminate. Clinical cure=resolution of acute signs, symptoms.Clinical improvement=participants switched to oral therapy;met following criteria at EOIV:afebrile for 24 hours(H);improvement in at least 1 symptom,sign.Clinical failure=received >48H of therapy, met any of these:therapy discontinuation due to insufficient effect, AE, death. Indeterminate=data not available for evaluation(death;lost to follow up;diagnosis of CNS infection, osteomyelitis, endocarditis or necrotizing enterocolitis after enrollment). EOIV (Up to 14 days), EOT (Up to 27 days), TOC (Up to 34 days), LFU (Up to 49 days).
Time Frame: EOIV, EOT, TOC, LFU
Population: ITT population set included all participants who had been enrolled in each part of the study, regardless of whether or not treatment was received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 8 | 5 | 8
Participants
  EOIV: Clinical cure | 2 | 2 | 3
  EOIV: Clinical improvement | 6 | 2 | 3
  EOIV: Clinical failure | 0 | 0 | 1
  EOIV: Indeterminate | 0 | 1 | 1
  EOIV: Missing | 0 | 0 | 0
  EOT: Clinical cure | 6 | 3 | 3
  EOT: Clinical improvement | 2 | 1 | 3
  EOT: Clinical failure | 0 | 0 | 1
  EOT: Indeterminate | 0 | 1 | 0
  EOT: Missing | 0 | 0 | 1
  LFU: Clinical cure | 8 | 4 | 6
  LFU: Clinical improvement | 0 | 0 | 0
  LFU: Clinical failure | 0 | 0 | 1
  LFU: Indeterminate | 0 | 1 | 0
  LFU: Missing | 0 | 0 | 0
  TOC: Clinical cure | 7 | 3 | 7
  TOC: Clinical improvement | 0 | 0 | 0
  TOC: Clinical failure | 0 | 0 | 1
  TOC: Indeterminate | 0 | 2 | 0
  TOC: Missing | 0 | 0 | 0

12. Secondary Outcome: Number of Participants According to Clinical Outcome At End of IV Treatment(EOIV), End of Treatment(EOT), Test of Cure(TOC) and Late Follow-Up(LFU) in Micro-ITT Analysis Population: Part B
Description: as for outcome 11
Time Frame: EOIV, EOT, TOC, LFU
Population: Micro ITT population included all participants who had at least 1 gram-negative pathogen in an adequate initial/prestudy culture. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 7 | 0 | 3
Participants
  EOIV: Clinical cure | 2 |  | 1
  EOIV: Clinical improvement | 5 |  | 0
  EOIV: Clinical failure | 0 |  | 1
  EOIV: Indeterminate | 0 |  | 1
  EOIV: Missing | 0 |  | 0
  EOT: Clinical cure | 6 |  | 1
  EOT: Clinical improvement | 1 |  | 0
  EOT: Clinical failure | 0 |  | 1
  EOT: Indeterminate | 0 |  | 0
  EOT: Missing | 0 |  | 1
  LFU: Clinical cure | 7 |  | 1
  LFU: Clinical improvement | 0 |  | 0
  LFU: Clinical failure | 0 |  | 1
  LFU: Indeterminate | 0 |  | 0
  LFU: Missing | 0 |  | 0
  TOC: Clinical cure | 6 |  | 2
  TOC: Clinical improvement | 0 |  | 0
  TOC: Clinical failure | 0 |  | 1
  TOC: Indeterminate | 0 |  | 0
  TOC: Missing | 0 |  | 0

13. Secondary Outcome: Number of Participants According to Clinical Outcome At End of IV Treatment(EOIV), End of Treatment(EOT), Test of Cure(TOC) and Late Follow-Up(LFU) in Modified-ITT Analysis Population: Part B
Description: as for outcome 11
Time Frame: EOIV, EOT, TOC, LFU
Population: Modified Intent-to-Treat (MITT) population included all participants who received any amount of CAZ-AVI and met minimal disease criteria of infection (defined as the presence of at least 1 clinical criterion and 1 laboratory criterion or met at least 2 clinical criteria in the presence of, or as a result of suspected or proven bacterial infection which required IV antibiotic therapy). Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 8 | 3 | 5
Participants
  EOIV: Clinical cure | 2 | 1 | 3
  EOIV: Clinical improvement | 6 | 1 | 0
  EOIV: Clinical failure | 0 | 0 | 1
  EOIV: Indeterminate | 0 | 1 | 1
  EOIV: Missing | 0 | 0 | 0
  EOT: Clinical cure | 6 | 1 | 3
  EOT: Clinical improvement | 2 | 1 | 0
  EOT: Clinical failure | 0 | 0 | 1
  EOT: Indeterminate | 0 | 1 | 0
  EOT: Missing | 0 | 0 | 1
  LFU: Clinical cure | 8 | 2 | 3
  LFU: Clinical improvement | 0 | 0 | 0
  LFU: Clinical failure | 0 | 0 | 1
  LFU: Indeterminate | 0 | 1 | 0
  LFU: Missing | 0 | 0 | 0
  TOC: Clinical cure | 7 | 1 | 4
  TOC: Clinical improvement | 0 | 0 | 0
  TOC: Clinical failure | 0 | 0 | 1
  TOC: Indeterminate | 0 | 2 | 0
  TOC: Missing | 0 | 0 | 0

14. Secondary Outcome: Number of Participants According to Microbiological Response at TOC Visit in Micro-ITT Population: Part B
Description: Microbiological response was assessed based on eradication, presumed eradication, persistence, presumed persistence, indeterminate. Eradication: source specimen demonstrated absence of the original baseline pathogen. Presumed eradication: source specimen was not available to culture and the participant was assessed as a clinical cure. Persistence: source specimen demonstrated continued presence of the original baseline pathogen. Presumed persistence: source specimen was not available to culture and the participant was assessed as a clinical failure. Indeterminate: source specimen was not available to culture and the participant's clinical outcome was assessed as indeterminate.
Time Frame: Up to 34 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 7 | 0 | 3
Participants
  Enterobacter Cloacae Complex: F: Eradication | 0 |  | 0
  Enterobacter Cloacae Complex: F: Presumed eradication | 0 |  | 0
  Enterobacter Cloacae Complex: U: Persistence | 0 |  | 0
  Enterobacter Cloacae Complex: U: Presumed persistence | 0 |  | 1
  Enterobacter Cloacae Complex Indeterminate | 0 |  | 0
  E.coli: F: Eradication | 4 |  | 0
  E.coli: F: Presumed eradication | 2 |  | 0
  E.coli: U: Persistence | 0 |  | 0
  E.coli:U:Presumed persistence | 0 |  | 0
  E.coli:Indeterminate | 0 |  | 0
  Klebsiella Oxytoca:F: Eradication | 0 |  | 0
  Klebsiella Oxytoca:F:Presumed eradication | 0 |  | 1
  Klebsiella Oxytoca:U: Persistence | 0 |  | 0
  Klebsiella Oxytoca:U:Presumed persistence | 0 |  | 0
  Klebsiella Oxytoca: Indeterminate | 0 |  | 0
  Klebsiella Pneumoniae:F: Eradication | 0 |  | 0
  Klebsiella Pneumoniae:F:Presumed eradication | 0 |  | 1
  Klebsiella Pneumoniae:U: Persistence | 0 |  | 0
  Klebsiella Pneumoniae:U:Presumed persistence | 0 |  | 0
  Klebsiella Pneumoniae: Indeterminate | 0 |  | 0

15. Secondary Outcome: Number of Participants With Emergent Infections in Micro-ITT Analysis Population: Part B
Description: Emergent infections included superinfection and new infection. Superinfection: a culture identified pathogen other than a baseline pathogen during the course of active treatment with study therapy requiring alternative antimicrobial therapy. New infection: a culture identified pathogen other than a baseline pathogen at any time after study treatment has finished requiring alternative antimicrobial therapy.
Time Frame: Day 1 up to maximum of Day 49
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 7 | 0 | 3
Participants
  Superinfection | 0 | 0 | 0
  New infection | 0 | 0 | 0

16. Primary Outcome: Number of Participants With Clinically Significant Laboratory Parameters Occurred in More Than 2 Participants: Part B
Description: Number of participants in Part B with clinically significant abnormal laboratory parameters that occurred in more than 2 participants from Day 1 up to 35 days after the last dose of CAZ-AVI were reported in this outcome measure. Clinically significant labs were abnormal laboratory results which the investigator reported as being clinically significant. Only parameters with non-zero values are reported.
Time Frame: Day 1 up to maximum of Day 49
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
Number analyzed (Participants) | 8 | 5 | 8
Participants
  Hematology: Hematocrit | 2 | 0 | 1
  Hematology: Hemoglobin | 2 | 0 | 2
  Hematology: Leukocytes | 0 | 2 | 1
  Hematology: Neutrophils/Leukocytes | 1 | 2 | 0
  Hematology: Platelets | 1 | 1 | 2
  Clinical Chemistry:Alanine Aminotransferase | 1 | 1 | 1
  Clinical Chemistry: Albumin | 1 | 2 | 2
  Clinical Chemistry: Aspartate Aminotransferase | 1 | 2 | 1
  Clinical Chemistry: Base Excess | 0 | 3 | 3
  Clinical Chemistry: Bilirubin | 0 | 1 | 2
  Clinical Chemistry: Blood Ph | 0 | 3 | 3
  Clinical Chemistry: C Reactive Protein | 2 | 4 | 8
  Clinical Chemistry: Direct Bilirubin | 0 | 1 | 3
  Clinical Chemistry:Partial Pressure Carbon Dioxide | 0 | 1 | 2
  Clinical Chemistry: Potassium | 0 | 2 | 1
  Clinical Chemistry: Procalcitonin | 0 | 2 | 4

17. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Parameters Occurred in More Than 2 Participants: Part A
Description: Number of participants in Part A with clinically significant abnormal laboratory parameters that occurred in more than 2 participants from Day 1 up to 35 days after the last dose of CAZ-AVI were reported in this outcome measure. Clinically significant labs were abnormal laboratory results which the investigator reported as being clinically significant.
Time Frame: Day 1 up to maximum of Day 35
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3
Number analyzed (Participants) | 9 | 8 | 8
Participants
  Hematology: Hematocrit | 1 | 1 | 2
  Hematology: Hemoglobin | 1 | 1 | 2
  Hematology: Leukocytes | 1 | 2 | 3
  Blood chemistry | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part A: Day 1 up to maximum of Day 35; Part B: Day 1 up to maximum of Day 49
Description: Same event may appear as both SAE and non-SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety Analysis Sets for Part A and Part B included participants who received any amount of the investigational drug (CAZ-AVI) in the respective part. The death reported in Part B: cohort 1 occurred after participant completed the study (including safety follow-up).
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3 | Part B: Cohort 1 | Part B: Cohort 2 | Part B: Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/8 | 0/8 | 0/5 | 1/8
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/8 | 1/8 | 1/8 | 2/5 | 2/8
Other Adverse Events (participants affected / at risk) | 1/9 | 0/8 | 1/8 | 3/8 | 1/5 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Cohort 1 (N=9) | Part A: Cohort 2 (N=8) | Part A: Cohort 3 (N=8) | Part B: Cohort 1 (N=8) | Part B: Cohort 2 (N=5) | Part B: Cohort 3 (N=8)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Necrotising colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Candida sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Cohort 1 (N=9) | Part A: Cohort 2 (N=8) | Part A: Cohort 3 (N=8) | Part B: Cohort 1 (N=8) | Part B: Cohort 2 (N=5) | Part B: Cohort 3 (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04126031/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT04126031/SAP_001.pdf